CLINICAL TRIAL: NCT03491709
Title: A Preliminary Clinical Study on the Pharmacokinetics and Safety of Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) in Patients With Advanced Colorectal Cancer or Head and Neck Squamous Cell Carcinoma
Brief Title: A Preliminary Clinical Study on the Pharmacokinetics and Safety of CDP1 in Patients With Advanced CRC or HNSCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDP100001
Record Dates: First submitted 2018-03-21; First posted 2018-04-09 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-EGFR monoclonal antibody (Experimental): Recombinant anti-EGFR human mouse chimeric monoclonal antibody injection 250mg/m2 single administration
  Interventions: Drug: anti-EGFR monoclonal antibody
- Cetuximab injection (Active Comparator): Cetuximab,Erbitux 250mg/m2 single administration
  Interventions: Drug: Cetuximab injection

INTERVENTIONS:
Drug: anti-EGFR monoclonal antibody — Recombinant anti-EGFR human mouse chimeric monoclonal antibody injection
  Other Names: CDP1
  Arms: anti-EGFR monoclonal antibody
Drug: Cetuximab injection — Cetuximab injection
  Other Names: Erbitux
  Arms: Cetuximab injection

SUMMARY:
Colorectal cancer (CRC) is one of the most common human malignant tumors. The incidence and mortality of colorectal cancer in our country are on the rise. Surgery-based, combined with chemotherapy, radiotherapy comprehensive treatment, is the main treatment of colorectal cancer. Surgical resection has been recognized as the primary treatment of colorectal cancer. However, due to the majority of patients already advanced at the time of diagnosis, some difficulties are brought to radical surgery. Therefore, the importance of chemotherapy for colorectal cancer gradually been clinically recognized, But rarely survive more than 18 months." In addition to chemotherapy, there is now a more ideal model of cancer treatment- molecular targeted therapies, including monoclonal antibody drugs such as cetuximab, as well as small molecule tyrosine kinases Inhibitors gefitinib and so on. Molecular targeted drugs make use of the difference in molecular biology between tumor cells and normal cells. Targeting drugs to tumor cells and inhibiting the growth and proliferation of the cells can achieve the therapeutic effect, which has the advantages of high specificity and low adverse reaction. The bio-targeted drug cetuximab is the first drug approved to marketed as an epidermal growth factor receptor (EGFR)-targeting immunoglobulin 1（IgG1）monoclonal antibody. Cetuximab, either monotherapy or combined radiotherapy and chemotherapy, can exert excellent anti-tumor activity in EGFR-positive malignant tumors and can significantly enhance the efficacy of radiotherapy and chemotherapy.

Reference to cetuximab injection, guilin sanjin Co., Ltd. and dragonboat Co., Ltd. jointly developed a recombinant anti-EGFR human mouse chimeric monoclonal antibody (R & D code: CDP1).The primary structure of CDP1 is exactly the same with cetuximab, the higher structure and Physical and chemical properties and cetuximab are highly similar. Pharmacodynamic activity in vivo and in vitro, pharmacokinetic characteristics and toxicological reactions are also similar to cetuximab. CDP1 selected with cetuximab consistent formulations, prescriptions, specifications.

CDP1 was approved by China Food and Drug Administration (No. 2016L06884) in August 2016 for clinical studies. According to the contents of the document and guidelines for biological analogs, the clinical pharmacokinetic and clinical effectiveness comparison tests of CDP1 and the safety and immunogenicity assessment are planned.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To compare the pharmacokinetic characteristics of a single dose between CDP1 and the original drug Erbitux In patients with advanced metastatic colorectal cancer.

Secondary :

1. To compare the safety and immunogenic characteristics of the single dose between CDP1 and the original drug Erbitux in patients with advanced metastatic colorectal cancer.
2. To evaluate the pharmacokinetics and safety of CDP1 multiple administrations."

OUTLINE

The study can be divided into 3 parts:

Part 1: Single-dose Phase:

single center, parallel, randomized, single-blind trial. The original drug Erbitux as a control, CDP1 and Erbitux single-dose pharmacokinetics of the initial comparison, and at the same time safety and immunogen preliminary comparison. CDP1 group received a single administration of CDP1 250mg/m2, Erbitux group received Erbitux 250mg/m2 single administration. Two groups of subjects after a single administration into the 4-week observation period, safety observations, pharmacokinetic blood samples and immunogenic blood samples were collected. The tumor was evaluated at the end of the 4 week observation period.If the subjects did not develop the disease, or did not appear the intolerant toxicity during the observation period, they entered the period of multiple drug delivery.

Part 2: Multi-dose Phase:

Single center, single arm, open trial, evaluation of pharmacokinetics and safety with multiple doses of CDP1. Multiple administrations of two groups of subjects were followed by continuous administration of CDP1. Dosing regimen is the first administration of 400mg/m2, followed by 250mg/m2, once a week for 6 weeks.

Part 3: Follow-up Phase:

CDP1, IV, once a week, 250mg/m2, until the patient's death or the withdrawal decision of the patient and/or investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 75 (inclusive) years , male.
* Histologically or cytologically confirmed ras genotype is wild-type patients with advanced metastatic colorectal cancer, at least second-line chemotherapy (including oxaliplatin, irinotecan and fluorouracil drugs) failed, or intolerant to Irinotecan or chemotherapy-denied patients.
* ECOG physical score 0-2 points.
* Expected survival time of 3 months or more.
* According to RECIST 1.1, there is at least one assessable tumor lesion.
* No serious hematological system, liver function, renal function and coagulation dysfunction:Neutrophils ≥1.5 × 109 / L, platelets ≥75 × 109 / L, hemoglobin≥90g / L; total bilirubin≤1.5 times ULN, alanine aminotransferase (ALT)≤2.5 times ULN,aspartate transaminase (AST) ≤2.5 times ULN (liver metastasis ALT ≤ 5 times ULN, AST≤ 5 times ULN);Serum creatinine ≤1.5 times ULN;Activated partial thromboplastin time (APTT) ≤1.5 times ULN, prothrombin time (PT) ≤1.5 times ULN, international normalized ratio (INR) ≤1.5 times ULN.
* Eligible patients with fertility must agree to use reliable methods of contraception (hormonal or barrier abstinence) for at least 12 weeks during and after the last dose of medication.
* Subjects should be informed of the study prior to the test and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Chemotherapy, biotherapy, radiation therapy, endocrine therapy, small molecule targeted therapies and other anti-tumor, etc. within 4 weeks prior to the start of study drug use or within 5 half-lives of the known drug (whichever is longer) Anti-cancer therapy, or other experimental drug treatment (except nitrosourea, mitomycin C and fluorouracil oral drugs),nitrosourea or mitomycin C for 6 weeks. Fluorouracil-based oral medications, such as tiotropium and capecitabine, have an interval of at least 2 weeks between the last oral dose and study drug use.
* Have previously received anti-EGFR monoclonal antibody treatment.
* EGFR antibody drug-resistant antibody (ADA) positive.
* Within 3 months prior to enrollment, major organ surgery (excluding biopsy) or significant trauma occurred.
* The adverse reactions of previous anti-tumor therapy have not been restored to CTCAE 4.03 grade ≤1 (excluding hair loss).
* Untreated or clinically symptomatic brain metastases, spinal cord compression, cancerous meningitis, or other evidence that the patient's brain, spinal metastases have not yet been controlled, the researchers judged not suitable for inclusion. clinical symptoms suspected brain or soft Membrane disease is to be ruled out by CT / MRI examination.
* Uncontrolled active infections.
* Have a history of immunodeficiency, including HIV antibody test positive.
* Treponema anti-positive.
* Chronic hepatitis B virus (HBV) infection; Hepatitis C virus (HCV) infection.
* Serious history of cardiovascular disease: including ventricular arrhythmias requiring clinical intervention; acute coronary syndromes, congestive heart failure, stroke or other cardiovascular events of grade III and higher within 6 months; New York, USA Heart Association (NYHA. Cardiac function grade ≥II or Left ventricular ejection fraction(LVEF) <50%; poorly controlled hypertension (systolic blood pressure> 150 mmHg, diastolic blood pressure> 90 mmHg).
* Interstitial lung disease.
* There are other serious history of systemic diseases, the researchers judged not suitable for clinical trials of patients.
* Alcohol or drug dependence is known.
* Persons with mental disorders or poor compliance.
* Moderate or severe infusion-related reactions, including anaphylaxis, have been reported in the past when using monoclonal antibody drugs.
* The investigators did not find it appropriate to participate in this clinical study because of any clinical or laboratory abnormalities or other causes.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Age 18 ~ 75 (inclusive) years , male
Enrollment: 18 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters: Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters: AUC(0-t) for CDP1

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-00) After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters: AUC(0-00) for CDP1
Pharmacokinetic parameters: Observed Maximum Serum Concentration (Cmax) of CDP1 After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters Cmax for CDP1
Pharmacokinetic parameters: Mean Residence Time of Drug in the Body (MRT) of CDP1 After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters MRT for CDP1
Pharmacokinetic parameters: Apparent Terminal Half-life (t1/2) of CDP1 After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters T1/2 for CDP1
Pharmacokinetic parameters: Total Body Clearance of Drug From Serum (CL) After First Infusion | Up to 59 Days
  Single-dose Phase: Pharmacokinetic parameters CL for CDP1
Vital signs: Blood pressure | Up to 73 Days
  Vital signs: Blood pressure
Vital signs: Pulse rate | Up to 73 Days
  Vital signs: Pulse rate
Vital signs: Respiratory rate | Up to 73 Days
  Vital signs: Respiratory rate
Physical examination: height | Up to 73 Days
  Physical examination: height
Physical examination: Weigh | Up to 73 Days
  Physical examination: Weigh
Number of Subjects With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score vs. Worst Post-baseline Score | Up to 73 Days
  ECOG performance status measured to assess subject's performance status on a scale of 0 to 4, where 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair. ECOG performance status was reported in terms of number of subjects with Baseline value vs. worst post-baseline value (i.e. highest score) combination.
Number of Subjects With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score vs. Best Post-baseline Score | Up to 73 Days
  ECOG performance status measured to assess subject's performance status on a scale of 0 to 4, where 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair. ECOG performance status was reported in terms of number of subjects with Baseline value vs. best post-baseline value (i.e. lowest score) combination.
Frequency of adverse events (AE) | Up to 59 Days
  Frequency of adverse events (AE)
Immunogenicity indicators: Anti-drug antibodies (ADA) . | Up to 73 Days
  Immunogenicity indicators: Anti-drug antibodies (ADA) .
Immunogenicity indicators: neutralizing antibodies | Up to 73 Days
  Immunogenicity indicators: neutralizing antibodies (Titers and Nab analyzes will be performed when ADA screening is positive).

CONTACTS AND LOCATIONS:
Overall Officials: Li Jin, doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital Phase 1 Clinical Trial Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No